CLINICAL TRIAL: NCT04122924
Title: Effect of Abdominal Muscle Training on Inter-recti Distance and Prevalence of Diastasis Recti Abdominis in Postpartum Primi- and Multiparous Women: A Randomized Controlled Trial
Brief Title: Postpartum Exercise and Diastasis Recti Abdominis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian School of Sport Sciences (Other)
Collaborators: The Norwegian Women´s Public Health Association (Other)
Responsible Party: Principal Investigator, Kari Bø, Prof, PhD, PT, Exercise scientist, Norwegian School of Sport Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SLG89
Record Dates: First submitted 2019-10-04; First posted 2019-10-10 (Actual); Last update posted 2023-03-02 (Actual); Status verified 2023-03

CONDITIONS: Diastasis Recti Abdominis; Diastasis Recti
Keywords: Postpartum; Abdominal Muscle Training; Exercise
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Intervention Model Description: An assessor blinded parallel group RCT
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): A three months home-based abdominal muscle training program.
  Interventions: Other: Abdominal muscle training
- Control Group (No Intervention): The control group will have no intervention, and will be asked not to attend any specific supervised abdominal muscle training program during the 3 months intervention period.

INTERVENTIONS:
Other: Abdominal muscle training — The intervention starts 6-12 months postpartum and will last for three months with weekly follow-up through an exercise app. Before commencing the home-based program, women in the intervention group will have an individual session in how to perform the program with a physiotherapist. The intervention consists of a 10 min 5 days a week exercise program, including the following exercises; headlift, crunch and twisted crunch. General principles for strength training are followed: 3 sets of 8-12 contractions close to maximum. The participants will be provided with a smartphone app (Athlete Monitoring) to be reminded to exercise and to register adherence.
  Arms: Intervention Group

SUMMARY:
Prevalence rates of diastasis recti abdominis (DRA) among postpartum women vary between 30% - 68%. It has been postulated that DRA, in addition to being a cosmetic concern for many women, may reduce low- back and pelvic stability causing low back- and pelvic girdle pain and be related to pelvic floor dysfunctions such as urinary incontinence, anal incontinence and pelvic organ prolapse. Given the limited research data, there is currently no consensus on which abdominal exercises to recommend to narrow the diastasis.

The purpose of this assessor blinded parallel group randomized controlled trial (RCT) is to evaluate the effect of abdominal muscle training on inter-recti distance (IRD) and prevalence of DRA.

DETAILED DESCRIPTION:
BACKGROUND:

DRA is defined as an impairment with midline separation of the two rectus abdominis muscles along the linea alba. The condition affects a significant number of women during the antenatal- and postnatal period. Today there is a strong focus on the pregnant woman's appearance, especially through social media. Webpages and apps recommend how women should stay thin and get back into shape with "a flat tummy" at an early stage of the postpartum period. There are easily available advices on how to get rid of what is named "the mum's belly" (e.g.mammamage.se, breakingmuscle.com, befitmom.com, babybellybelt.com, tummyzip.com). A systematic review of the scientific literature has found none or very weak evidence behind any of these advices. DRA is diagnosed by measuring the distance between the median borders of the two rectus abdominis; IRD, and ultrasound has been found to have the best intra- and inter-tester reliability with Intraclass Correlation Coefficient (ICC) > 0.9.

In a systematic review by Benjamin et al. (2014), 8 studies in treatment of DRA using abdominal exercises were found: four case studies, two retrospective observational studies, one quasi-experimental post-test study and one small RCT of a brief training intervention. A new search on Pubmed of July 2019 found six additional RCTs using abdominal exercises in treatment of DRA. The studies differ in methodological and interventional quality and results differ between studies. Given the limited research data, use of different outcome measures and cut-off point for diastasis in published studies, there is currently no consensus on which abdominal exercises to recommend to narrow the diastasis.

AIMS:

The aim of this study is to assess the effect of abdominal muscle training on IRD and prevalence of DRA in postpartum primi- and multiparous women.

STUDY DESIGN AND METHODS:

Before starting this RCT, an experimental cross-sectional study investigating the acute effect of different abdominal- and pelvic floor exercises on IRD in women with DRA will be conducted. Based on findings from the experimental cross-sectional study, we will choose exercises that narrow the IRD for the RCT's exercise program.

Women will respond to an electronic questionnaire sent by email before they meet for the clinical assessments, before and after the intervention period. Women diagnosed with DRA giving informed consent are assessed at baseline with 2D ultrasound measurements of IRD, abdominal muscle strength tests and the Oswestry Low Back Disability Index (ODI), Pelvic Girdle Questionnaire (PGQ) and (Pelvic Floor Disability Index) PFDI-20. After baseline testing the participants are randomly allocated to either an exercise or control group. Randomization will be computer-generated, in blocks of 4 with concealed allocation. Randomization will be provided by a person not involved in assessments of outcome. The outcome assessor will be blinded for group allocation. After the 3 month training period, both the exercise and control group will be reassessed with 2D ultrasound, abdominal muscle strength and endurance tests and the ODI, PGQ and PFDI-20.

ELIGIBILITY:
Inclusion Criteria:

* Primi- and multiparous women 6-12 months postpartum
* Understand instructions given in Norwegian language
* Willing/available to participate in a 3 months intervention period

Exclusion Criteria:

* Pregnant women
* Women < 6 months or > 12 months postpartum
* Women with children with illnesses and mothers with neurological, systemic musculoskeletal diseases or psychiatric diagnoses will be excluded from participation
* Women with adherence < 70 % of the home-based program will be excluded for the per protocol analyzes
* Women with specific need for pelvic floor muscle training during the 3 months intervention period will be excluded

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 70 (Actual)
Dates: Start 2020-01-09 (Actual); Primary Completion 2022-12-21 (Actual); Study Completion 2022-12-21 (Actual)

PRIMARY OUTCOMES:
Change in IRD assessed by 2D ultrasonography | Change from baseline IRD at 3 months
  A portable 2D ultrasound (GE Healthcare -Logiq e R7) will be used to assess IRD inn mm at 2 cm above and 2 cm below (P. G. Mota et al., 2015a) the umbilicus during rest and crunch.

SECONDARY OUTCOMES:
Change in abdominal endurance | Change from baseline abdominal endurance at 3 months
  Abdominal endurance will be assessed as number of repetitions of one standardized abdominal crunch to exhaustion (ACSM, 2006).
Change in abdominal strength | Change from baseline abdominal strength at 3 months
  Maximal abdominal strength will be measured in a trunk dynamometer (HUMAC NORM).
Change in cross-sectional area of m. rectus abdominis | Change from baseline cross-sectional area at 3 months
  Cross-sectional area of m. rectus abdominis will be measured by 2D ultrasonography, above and below the umbilicus.
Change in symptoms of low back pain | Change from baseline symptoms of low back pain at 3 months
  The electronic questionnaires include the following instrument: Oswestry Low Back Disability Index (ODI).
Change in symptoms of pelvic girdle pain | Change from baseline symptoms of pelvic girdle pain at 3 months
  The electronic questionnaire include the following instrument: Pelvic Girdle Questionnaire (PGQ).
Change in symptoms of pelvic floor dysfunctions | Change from baseline symptoms of pelvic floor dysfunctions at 3 months
  The electronic questionnaire include the following instrument: Pelvic Floor Disability Index (PFDI-20).
Global rating of change (GRC) | Post-test after a 3-months intervention period
  Perceived change of the condition will be assessed by a numerical 11-point scale. A 11-point scale with response choices ranging from "completely recovered" to "very much worse".

CONTACTS AND LOCATIONS:
Overall Officials: Kari Bø, PhD, Study Chair — Norwegian School of Sport Sciences
Locations (1):
- Norwegian School of Sport Sciences, Department of Sports Medicine, Oslo, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rett, M. T., Braga, M., Bernardes, N., & Andrade, S. (2009). Prevalence of diastasis of the rectus abdominis muscles immediately postpartum: comparison between primiparae and multiparae. Revista Brasileira De Fisioterapia, 13(4), 275-280. doi:10.1590/s1413-35552009005000037
- [Background] Turan V, Colluoglu C, Turkyilmaz E, Korucuoglu U. Prevalence of diastasis recti abdominis in the population of young multiparous adults in Turkey. Ginekol Pol. 2011 Nov;82(11):817-21. PMID 22384613
- [Background] Lee DG, Lee LJ, McLaughlin L. Stability, continence and breathing: the role of fascia following pregnancy and delivery. J Bodyw Mov Ther. 2008 Oct;12(4):333-48. doi: 10.1016/j.jbmt.2008.05.003. Epub 2008 Jul 1. PMID 19083692
- [Background] Spitznagle TM, Leong FC, Van Dillen LR. Prevalence of diastasis recti abdominis in a urogynecological patient population. Int Urogynecol J Pelvic Floor Dysfunct. 2007 Mar;18(3):321-8. doi: 10.1007/s00192-006-0143-5. Epub 2006 Jul 26. PMID 16868659
- [Background] Venes, D., & Taber, C. (2013). Taber's cyclopedic medical dictionary (22. ed.). Philadelphia: FA Davis Co
- [Background] Benjamin DR, van de Water AT, Peiris CL. Effects of exercise on diastasis of the rectus abdominis muscle in the antenatal and postnatal periods: a systematic review. Physiotherapy. 2014 Mar;100(1):1-8. doi: 10.1016/j.physio.2013.08.005. Epub 2013 Oct 5. PMID 24268942
- [Background] Mota P, Pascoal AG, Sancho F, Bo K. Test-retest and intrarater reliability of 2-dimensional ultrasound measurements of distance between rectus abdominis in women. J Orthop Sports Phys Ther. 2012 Nov;42(11):940-6. doi: 10.2519/jospt.2012.4115. Epub 2012 Jul 18. PMID 22810966
- [Background] Mesquita, L. A., Machado, A. V., & Andrade, A. V. (1999). Physiotherapy for reduction of diastasis of the recti adbominis muscles in the postpartum period. Rev Brasil Ginecol Obstet 21, 267-272.
- [Background] Emanuelsson P, Gunnarsson U, Dahlstrand U, Strigard K, Stark B. Operative correction of abdominal rectus diastasis (ARD) reduces pain and improves abdominal wall muscle strength: A randomized, prospective trial comparing retromuscular mesh repair to double-row, self-retaining sutures. Surgery. 2016 Nov;160(5):1367-1375. doi: 10.1016/j.surg.2016.05.035. Epub 2016 Jul 27. PMID 27475817
- [Background] Gluppe SL, Hilde G, Tennfjord MK, Engh ME, Bo K. Effect of a Postpartum Training Program on the Prevalence of Diastasis Recti Abdominis in Postpartum Primiparous Women: A Randomized Controlled Trial. Phys Ther. 2018 Apr 1;98(4):260-268. doi: 10.1093/ptj/pzy008. PMID 29351646
- [Background] Kamel DM, Yousif AM. Neuromuscular Electrical Stimulation and Strength Recovery of Postnatal Diastasis Recti Abdominis Muscles. Ann Rehabil Med. 2017 Jun;41(3):465-474. doi: 10.5535/arm.2017.41.3.465. Epub 2017 Jun 29. PMID 28758085
- [Background] Tuttle, L. J., Fasching, J., Keller, A., Patel, M., Saville, C., Schlaff, R., . . . Gombatto, S. P. (2018). Noninvasive Treatment of Postpartum Diastasis Recti Abdominis: A Pilot Study. Journal of Women's Health Physical Therapy, 42(2), 65-75. doi:10.1097/jwh.0000000000000101
- [Background] Walton, L. M., Costa, A., LaVanture, D., McIlrath, S., & Stebbins, B. (2016). The effects of a 6 week dynamic core stability plank exercise program compared to a traditional supine core stability strengthening program on diastasis recti abdominis closure, pain, oswestry disability index (ODI) and pelvic floor disability index scores (PFDI). Physical Therapy and Rehabilitation, 3(1), 3. doi:10.7243/2055-2386-3-3
- [Background] Thabet AA, Alshehri MA. Efficacy of deep core stability exercise program in postpartum women with diastasis recti abdominis: a randomised controlled trial. J Musculoskelet Neuronal Interact. 2019 Mar 1;19(1):62-68. PMID 30839304
- [Background] Haskell WL, Lee IM, Pate RR, Powell KE, Blair SN, Franklin BA, Macera CA, Heath GW, Thompson PD, Bauman A; American College of Sports Medicine; American Heart Association. Physical activity and public health: updated recommendation for adults from the American College of Sports Medicine and the American Heart Association. Circulation. 2007 Aug 28;116(9):1081-93. doi: 10.1161/CIRCULATIONAHA.107.185649. Epub 2007 Aug 1. PMID 17671237
- [Background] Bø, K., et al. (1990). Pelvic floor muscle exercise for the treatment of female stress urinary incontinence: III. Effects of two different degrees of pelvic floor muscle exercises. Neurourol Urodyn 9(5): 489-502.
- [Background] Fairbank JC, Pynsent PB. The Oswestry Disability Index. Spine (Phila Pa 1976). 2000 Nov 15;25(22):2940-52; discussion 2952. doi: 10.1097/00007632-200011150-00017. PMID 11074683
- [Background] Stuge B, Garratt A, Krogstad Jenssen H, Grotle M. The pelvic girdle questionnaire: a condition-specific instrument for assessing activity limitations and symptoms in people with pelvic girdle pain. Phys Ther. 2011 Jul;91(7):1096-108. doi: 10.2522/ptj.20100357. Epub 2011 May 19. PMID 21596959
- [Background] Teig CJ, Grotle M, Bond MJ, Prinsen CAC, Engh MAE, Cvancarova MS, Kjollesdal M, Martini A. Norwegian translation, and validation, of the Pelvic Floor Distress Inventory (PFDI-20) and the Pelvic Floor Impact Questionnaire (PFIQ-7). Int Urogynecol J. 2017 Jul;28(7):1005-1017. doi: 10.1007/s00192-016-3209-z. Epub 2017 Jan 6. PMID 28062903
- [Background] Kamper SJ, Maher CG, Mackay G. Global rating of change scales: a review of strengths and weaknesses and considerations for design. J Man Manip Ther. 2009;17(3):163-70. doi: 10.1179/jmt.2009.17.3.163. PMID 20046623
- [Derived] Gluppe SB, Ellstrom Engh M, Bo K. Curl-up exercises improve abdominal muscle strength without worsening inter-recti distance in women with diastasis recti abdominis postpartum: a randomised controlled trial. J Physiother. 2023 Jul;69(3):160-167. doi: 10.1016/j.jphys.2023.05.017. Epub 2023 Jun 5. PMID 37286390